CLINICAL TRIAL: NCT01075854
Title: A Prospective, Multi-center, Observational Study of Gonal-F Filled by Mass Pens in Multifollicular Stimulation Prior to IVF/ICSI
Brief Title: An Observational Study of Gonal-F Filled by Mass Pens in Multifollicular Stimulation Prior to In-vitro Fertilization (IVF) or Intracytoplasmic Sperm Injection (ICSI)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Head of Medical Department, Merck Serono Korea, an affiliate of Merck KGaA, Darmstadt, Germany
Other Study IDs: EMR 700623_507
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2010-09

CONDITIONS: Multifollicular Stimulation
Keywords: Gonal-F; Multifollicular stimulation; Pregnancy; Ovarian hyperstimulation; In vitro fertilization; Intracytoplasmic sperm injection; Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples

INTERVENTIONS:
Drug: Gonal-F (Follitropin alfa) — Follitropin alfa FbM solution for injection in a prefilled pen is available in three strengths: 300 IU/0.5 ml (22 µg/0.5 ml), 450 IU/0.75 ml (33 µg/0.75 ml) and 900 IU/1.5 ml (66 µg/1.5 ml). The starting dose is usually recommended to be between 150 and 300 IU. The dose is then adjusted according to the ovarian response.
  Other Names: Gonal-F

SUMMARY:
This is a prospective, observational study in women using Gonal-F filled-by-mass (FbM) in ovarian hyperstimulation as part of their in-vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) treatment at infertility clinics in Korea. The purpose of this study is to assess Gonal-F FbM in a practical setting encompassing all subject groups and local practices.

DETAILED DESCRIPTION:
Follicle stimulating hormone (FSH) is a complex hetero-dimeric glycoprotein used therapeutically to stimulate follicular development in the ovary. The technical advance of recombinant technology to manufacture FSH has resulted in a biochemically pure FSH preparation with high batch-to-batch consistency. The protein content can be reliably quantified in mass units by size exclusion high performance liquid chromatography. These developments have enabled recombinant human FSH follitropin alfa (Gonal-F) to be filled and released in vials on the basis of mass with a variability of only ±2%. In one study, the FbM batches appeared to deliver a more consistent therapeutic effect than the filled-by-bioassay batches. In another randomized trial, self-administration and subjects' satisfaction were significantly higher in the pen device group than the conventional syringe group. Local reactions at injection sites and pain were significantly higher in the conventional syringe group than in the pen device group. The authors concluded that the pen device of Gonal-F is safe, convenient, and less painful, with more subject satisfaction than the conventional syringe form.

This prospective, multicentric, observational study is planned in women using Gonal-F FbM in ovarian hyperstimulation as part of their IVF/ICSI treatment at infertility clinics in Korea. Subjects fulfilling the eligibility criteria shall be enrolled in a consecutive manner over a 9-month period (approximately 1500 subjects).

OBJECTIVES

Primary objective:

* To assess the effectiveness Gonal-F FbM

Secondary objectives:

* To assess the safety and subject convenience of Gonal-F FbM in a normal clinical practice over a period of 9 months

ELIGIBILITY:
Inclusion Criteria:

* Women who are prescribed Gonal-F FbM by their treating physician for their IVF/ICSI treatment cycle will be eligible for this study

Exclusion Criteria:

* Subjects who have hypersensitivity to follitropin alfa, FSH or to any of the excipients
* Subjects with tumors of the hypothalamus and pituitary gland
* Ovarian enlargement or cyst not due to polycystic ovarian disease
* Gynecological hemorrhages of unknown etiology
* Ovarian, uterine or mammary carcinoma
* Primary ovarian failure
* Malformations of sexual organs incompatible with pregnancy
* Fibroid tumors of the uterus incompatible with pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female subjects who are prescribed Gonal-F FbM by their treating physician for their IVF/ICSI treatment cycle will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1539 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | Start of treatment to confirmation of pregnancy
  Number of oocytes retrieved and clinical pregnancy rate per cycle

SECONDARY OUTCOMES:
Efficacy, Safety and Convenience | Start of treatment to confirmation of pregnancy
  Secondary efficacy parameters includes total Gonal-f dose; stimulation profile of IVF cycle; number of follicles > 14 mm on day of hCG; number of available embryos; pregnancy status (hCG test, ultrasound exam); on the day of embryo transfer (ET).
  Convenience and safety parameters includes subject convenience rated by completing a questionnaire, local tolerance assessment (local reactions at the injection site, pain, satisfaction and convenience)

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Fertility Hospital, Seoul, South Korea